CLINICAL TRIAL: NCT01366898
Title: PROTOCOL FOR THE TREATMENT Acute Lymphoblastic Leukemia With Ph 'NEGATIVE IN ELDERLY PATIENTS (> 55 Years)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: PETHEMA Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LAL-07OLD
Record Dates: First submitted 2011-06-02; First posted 2011-06-06 (Estimated); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Idarubicin; Cytarabine; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Chemotherapy (Experimental)
  Interventions: Drug: Dexamethasona, Idarubicine, ARA-C, Methotrexate

INTERVENTIONS:
Drug: Dexamethasona, Idarubicine, ARA-C, Methotrexate

SUMMARY:
The protocol objective is providing adequate treatment and based on broad consensus in elderly patients with Acute Lymphoblastic Leukemia (ALL). Apply uniform treatment that enables a joint analysis of results strong enough to make conclusions on specific subgroups of patients (genotypic subtypes, particularly LAL Bcr/abl positive, phenotype, or strata of age or associated diseases). Provide results of a treatment to consider standard against which to compare the results of phase II trials of experimental drugs that undoubtedly will be activated in the coming years

DETAILED DESCRIPTION:
Prephase (days -5 to -1) Dexamethasone 10 mg/m2 bolus day IV for 5 days (-5 to -1). Supplementary treatment: hydration minimum 2000 ml/day, allopurinol 300 mg / day, gastric protection (as center), daily monitoring of blood glucose, daily monitoring of renal function. Intrathecal treatment (diagnosis and prophylactic) day -5: 12 mg were administered intrathecal methotrexate. The morphological study of the CSF will be defining initial CNS involvement by LAL. Although it is recommended immunophenotypic study of CSF, the definition of CNS involvement by LAL (and its therapeutic consequences) based on morphological observation of blasts in CSF cytocentrifuge.

Remission induction:

Tolerance prephase period can be used to establish the final indication of treatment (standard protocol or frail patients). Day 0 is free of treatment and is considered as +1 the first day of induction. The total duration of the induction is 30 days, consists of two phases (Phase I, days +1 to +14 and phase II, days +15 to +30). Mandatory testing is considered counting the percentage of blasts in peripheral blood +8 day of induction, a myelogram to day +14 to assess early response and a day +35 to assess the complete remission

(days +1 to +14)

* Vincristine (VCR) 1 mg (absolute dose) IV 1 and 8.
* Idarubicin (IDA): 10 mg (absolute dose) IV 1, 2, 8 and 9.
* Dexamethasone (DEX): 10 mg/m2 bolus days 1 and 2 IV, 8 to 11

days +15 to +30)

* cyclophosphamide (CFM): 300 mg / m 2 iV in 1 hour 15 to 17. (3 total doses).
* Cytarabine (ARAC): 60 mg / m 2 iV in 1 hour 16 to 19, 23 to 26. (8 total doses).
* Vincristine (VCR) 1 mg (absolute dose) iV 1 and 8.
* Idarubicin (IDA): 10 mg (absolute dose) iV 1, 2, 8 and 9.
* Dexamethasone (DEX): 10 mg/m2 bolus days 1 and 2 iV, 8 to 11

Consolidation:

Cycles 1, 3, 5 MTX: 1,000 mg/m2, IV infusion of 24 hours day 1 L-ASA. 10,000 IU / m 2 IV or IM Day 2 Cycles 2, 4, 6 ARAC: 1,000 mg/m2, IV in 3 hours on days 1, 3 and 5

ELIGIBILITY:
Inclusion Criteria:

Adults over 55 years diagnosed with ALL with chromosome Ph 'negative and naïve

Exclusion Criteria:

1. L3 ALL with mature B phenotype or cytogenetic abnormalities ALL characteristics of Burkitt type (t [8, 14], t [2, 8], t [8, 22]).
2. Biphenotypic acute leukemias and bilinear
3. Acute undifferentiated leukemia

   The criteria for exclusion from treatment (but not patient record) any of the following:
4. Patients with a history of severe and uncontrolled disease, including:

   * Coronary artery disease, valvular or hypertensive heart disease.
   * Chronic liver disease (active viral or alcoholic).
   * Chronic respiratory failure.
   * Renal failure not due to the ALL.
   * Serious neurological disorder not due to the ALL. f. Improperly controlled diabetes.
5. General condition affected (grades 3 and 4 of the WHO scale, see Appendix II), not attributable to the LAL.
6. LAL chromosome Ph 'positive (must register even if you follow a specific protocol).
7. Lack of consent by the patient to use their medical records.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2007-06-30 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy in terms of response rate | 5 years

SECONDARY OUTCOMES:
Efficacy in terms disease free survival | 5 years
Efficacy in terms of global survival | 10 years

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Germans Trias i Pujol and all Hospital Pethema, Badalona, Barcelona, Spain

REFERENCES:
- [Derived] Ribera JM, Garcia O, Fernandez-Abellan P, Lavilla E, Bernal MT, Gonzalez-Campos J, Brunet S, Monteserin MC, Montesinos P, Sarra J, Calbacho M, Alvarez-Larran A, Tormo M, Oriol A; PETHEMA Group. Lack of negative impact of Philadelphia chromosome in older patients with acute lymphoblastic leukaemia in the thyrosine kinase inhibitor era: comparison of two prospective parallel protocols. Br J Haematol. 2012 Nov;159(4):485-8. doi: 10.1111/bjh.12043. Epub 2012 Sep 12. No abstract available. PMID 22966847
- See also: Related Info — https://www.fundacionpethema.es/